CLINICAL TRIAL: NCT04944277
Title: Assessing Effectiveness of a Text-based Mental Health Coaching Application in Improving Mental Well-Being Among House Officers, IMU Faculty, IMU Corporate Staff and IMU Students in Malaysia
Brief Title: Assessing Effectiveness of ThoughtFullChat Application in Improving Mental Well-Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IMU University, Malaysia (Other)
Collaborators: ThoughtFull World Pte. Ltd. (Other)
Responsible Party: Principal Investigator, Lim Kean Ghee, Professor, IMU University, Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSc/Sem6(03)2021
Record Dates: First submitted 2021-06-10; First posted 2021-06-29 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Anxiety; Depression; Stress; Resilience
Keywords: Mental Health Wellbeing; Text-based Mental Health Coaching Application
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Without ThoughtFullChat Application (No Intervention): Participants will not use the app during the 3 months
- With ThoughtFullChat Application (Experimental): Participants will be using the app during the 3 months
  Interventions: Other: ThoughtFullChat Application

INTERVENTIONS:
Other: ThoughtFullChat Application — A subscription-based mobile platform that empowers users to proactively engage with their mental health via self-serve tools and 1-on-1 daily bite-sized coaching with certified mental health professionals.
  Arms: With ThoughtFullChat Application

SUMMARY:
* To determine the state of mental health among house officers, IMU corporate staff, IMU students and IMU faculty
* To find out the effectiveness and user experience of text-based mental health coaching applications among house officers, IMU corporate staff, IMU students and IMU faculty

IMU - International Medical University

DETAILED DESCRIPTION:
The text-based mental health coaching application that the investigators are using is ThoughtFullChat Application. ThoughtFullChat Application provides mental health coaching through text by licensed mental health professionals. Participants of this research will be required to answer a set of questionnaires which consists of DASS-21, Satisfaction with Life Scale and Brief Resilience Scale at the start of the study. Participants will be randomly distributed into 2 groups which are intervention and control groups. Participants in the intervention group will be using the application for 3 months. Post-intervention questionnaires will be given to all participants after 3 months. Data collected from these 2 groups will be analyzed by using SPSS.

ELIGIBILITY:
Inclusion Criteria:

* House Officers in Malaysia (UD41)
* Corporate staff in IMU, IMU Faculty Members
* All students who are currently studying in IMU who give their consent
* Competent in English Language
* Experiencing none to severe stress, anxiety or depression based on DASS-21 score

Exclusion Criteria:

* Medical students, Medical Officers (UD44)
* Contract staff, Outsourced staff or international staff in IMU campuses
* Students who refuse to give their consent and those that have already or just graduated from IMU
* Competent in other languages except English
* Experiencing extremely severe stress, anxiety or depression based on the DASS-21 score

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Anxiety | 3 months
  Depression, Anxiety and Stress Scale - 21 Items (DASS-21), a self report scale is used to measure the participants' emotional states of depression, anxiety and stress. For anxiety component, it contains 7 items and scores from 0 to 3 for each item. The total scores of each subscale need to be multiplied by 2 and are categorized into 5 severity ranges: normal, mild, moderate, severe and extremely severe. The severity ranges for anxiety are: normal (0-7); mild (8-9); moderate (10-14); severe (15-19) and extremely severe (20+).

SECONDARY OUTCOMES:
Depression | 3 months
  Depression, Anxiety and Stress Scale - 21 Items (DASS-21), a self report scale is used to measure the participants' emotional states of depression, anxiety and stress. For depression component, it contains 7 items and scores from 0 to 3 for each item. The total scores of each subscale need to be multiplied by 2 and are categorized into 5 severity ranges: normal, mild, moderate, severe and extremely severe. The severity ranges for depression are: normal (0-9); mild (10-13); moderate (14-20); severe (21-27) and extremely severe (28+).
Stress | 3 months
  Depression, Anxiety and Stress Scale - 21 Items (DASS-21), a self report scale is used to measure the participants' emotional states of depression, anxiety and stress. For stress component, it contains 7 items and scores from 0 to 3 for each item. The total scores of each subscale need to be multiplied by 2 and are categorized into 5 severity ranges: normal, mild, moderate, severe and extremely severe. The severity ranges for stress are: normal (0-14); mild (15-18); moderate (1-25); severe (26-33) and extremely severe (34+).
Resilience | 3 months
  Brief Resilience Scale is created to assess the perceived ability to bounce back or recover from stress. The scale was developed to assess a unitary construct of resilience, including both positively and negatively worded items. It consists of 6 items, each item scores from 1 to 5. Items 1, 3, 5 are positively worded while items 2, 4, 6 are negatively worded. The total score of Brief Resilience Scale will be the mean of the 6 items. The average score can be interpreted as follows: 1.00 to 2.99 (low resilience); 2.00 to 4.3 (normal resilience) and 4.31 to 5.00 (high resilience).
Satisfaction with Life | 3 months
  Satisfaction with Life Scale is developed to assess satisfaction with people's lives as a whole. The scale has 5 items with each item ranges from 1 to 7. The total range of scores is 5-35 while 20 point is the neutral point in the scale. The scores can be interpreted as follows: 5-9 (extremely dissatisfied with life), 31-35 (extremely satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Kean Ghee Lim, FRCS, Principal Investigator — International MU
Locations (1):
- IMU Clinical Campus, Seremban, Negeri Sembilan, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khan TM, Sulaiman SA, Hassali MA. Mental health literacy towards depression among non-medical students at a Malaysian university. Ment Health Fam Med. 2010 Mar;7(1):27-35. PMID 22477920
- [Background] Marshall JM, Dunstan DA, Bartik W. Effectiveness of Using Mental Health Mobile Apps as Digital Antidepressants for Reducing Anxiety and Depression: Protocol for a Multiple Baseline Across-Individuals Design. JMIR Res Protoc. 2020 Jul 5;9(7):e17159. doi: 10.2196/17159. PMID 32623368
- [Background] Kelders SM, Bohlmeijer ET, Pots WT, van Gemert-Pijnen JE. Comparing human and automated support for depression: Fractional factorial randomized controlled trial. Behav Res Ther. 2015 Sep;72:72-80. doi: 10.1016/j.brat.2015.06.014. Epub 2015 Jul 6. PMID 26196078
- [Background] Haider II, Tiwana F, Tahir SM. Impact of the COVID-19 Pandemic on Adult Mental Health. Pak J Med Sci. 2020 May;36(COVID19-S4):S90-S94. doi: 10.12669/pjms.36.COVID19-S4.2756. PMID 32582321
- [Background] Donker T, Petrie K, Proudfoot J, Clarke J, Birch MR, Christensen H. Smartphones for smarter delivery of mental health programs: a systematic review. J Med Internet Res. 2013 Nov 15;15(11):e247. doi: 10.2196/jmir.2791. PMID 24240579
- [Background] Hoyt R, Adler K, Ziesemer B, Palombo G. Evaluating the usability of a free electronic health record for training. Perspect Health Inf Manag. 2013 Apr 1;10(Spring):1b. Print 2013. PMID 23805062
- [Background] Teo AR, Choi H, Andrea SB, Valenstein M, Newsom JT, Dobscha SK, Zivin K. Does Mode of Contact with Different Types of Social Relationships Predict Depression in Older Adults? Evidence from a Nationally Representative Survey. J Am Geriatr Soc. 2015 Oct;63(10):2014-22. doi: 10.1111/jgs.13667. Epub 2015 Oct 6. PMID 26437566
- [Background] Abdul Latiff L, Tajik E, Ibrahim N, Abubakar AS, Ali SS. DEPRESSION AND ITS ASSOCIATED FACTORS AMONG SECONDARY SCHOOL STUDENTS IN MALAYSIA. Southeast Asian J Trop Med Public Health. 2016 Jan;47(1):131-41. PMID 27086434
- [Background] Adlina S, Suthahar A, Ramli M, Edariah AB, Soe SA, Mohd Ariff F, Narimah AH, Nuraliza AS, Karuthan C. Pilot study on depression among secondary school students in Selangor. Med J Malaysia. 2007 Aug;62(3):218-22. PMID 18246911
- [Background] Shamsuddin K, Fadzil F, Ismail WS, Shah SA, Omar K, Muhammad NA, Jaffar A, Ismail A, Mahadevan R. Correlates of depression, anxiety and stress among Malaysian university students. Asian J Psychiatr. 2013 Aug;6(4):318-23. doi: 10.1016/j.ajp.2013.01.014. Epub 2013 Mar 1. PMID 23810140
- [Background] Auerbach RP, Mortier P, Bruffaerts R, Alonso J, Benjet C, Cuijpers P, Demyttenaere K, Ebert DD, Green JG, Hasking P, Murray E, Nock MK, Pinder-Amaker S, Sampson NA, Stein DJ, Vilagut G, Zaslavsky AM, Kessler RC; WHO WMH-ICS Collaborators. WHO World Mental Health Surveys International College Student Project: Prevalence and distribution of mental disorders. J Abnorm Psychol. 2018 Oct;127(7):623-638. doi: 10.1037/abn0000362. Epub 2018 Sep 13. PMID 30211576
- [Background] Abdulghani HM, AlKanhal AA, Mahmoud ES, Ponnamperuma GG, Alfaris EA. Stress and its effects on medical students: a cross-sectional study at a college of medicine in Saudi Arabia. J Health Popul Nutr. 2011 Oct;29(5):516-22. doi: 10.3329/jhpn.v29i5.8906. PMID 22106758
- [Background] Dahlin M, Joneborg N, Runeson B. Stress and depression among medical students: a cross-sectional study. Med Educ. 2005 Jun;39(6):594-604. doi: 10.1111/j.1365-2929.2005.02176.x. PMID 15910436
- [Background] Hardeman RR, Przedworski JM, Burke SE, Burgess DJ, Phelan SM, Dovidio JF, Nelson D, Rockwood T, van Ryn M. Mental Well-Being in First Year Medical Students: A Comparison by Race and Gender: A Report from the Medical Student CHANGE Study. J Racial Ethn Health Disparities. 2015 Sep;2(3):403-13. doi: 10.1007/s40615-015-0087-x. PMID 26413458
- [Background] Jafari N, Loghmani A, Montazeri A. Mental health of Medical Students in Different Levels of Training. Int J Prev Med. 2012 Mar;3(Suppl 1):S107-12. PMID 22826751
- [Background] Puthran R, Zhang MW, Tam WW, Ho RC. Prevalence of depression amongst medical students: a meta-analysis. Med Educ. 2016 Apr;50(4):456-68. doi: 10.1111/medu.12962. PMID 26995484
- [Background] Patel V, Flisher AJ, Hetrick S, McGorry P. Mental health of young people: a global public-health challenge. Lancet. 2007 Apr 14;369(9569):1302-1313. doi: 10.1016/S0140-6736(07)60368-7. PMID 17434406
- [Background] Boyd CP, Hayes L, Nurse S, Aisbett DL, Francis K, Newnham K, Sewell J. Preferences and intention of rural adolescents toward seeking help for mental health problems. Rural Remote Health. 2011;11(1):1582. Epub 2011 Feb 14. PMID 21319934
- [Background] Arnett JJ. Emerging adulthood. A theory of development from the late teens through the twenties. Am Psychol. 2000 May;55(5):469-80. PMID 10842426
- [Background] Aysan F, Thompson D, Hamarat E. Test anxiety, coping strategies, and perceived health in a group of high school students: a Turkish sample. J Genet Psychol. 2001 Dec;162(4):402-11. doi: 10.1080/00221320109597492. PMID 11831350
- [Background] Bangasser DA, Curtis A, Reyes BA, Bethea TT, Parastatidis I, Ischiropoulos H, Van Bockstaele EJ, Valentino RJ. Sex differences in corticotropin-releasing factor receptor signaling and trafficking: potential role in female vulnerability to stress-related psychopathology. Mol Psychiatry. 2010 Sep;15(9):877, 896-904. doi: 10.1038/mp.2010.66. Epub 2010 Jun 15. PMID 20548297
- [Background] Bayram N, Bilgel N. The prevalence and socio-demographic correlations of depression, anxiety and stress among a group of university students. Soc Psychiatry Psychiatr Epidemiol. 2008 Aug;43(8):667-72. doi: 10.1007/s00127-008-0345-x. Epub 2008 Apr 8. PMID 18398558
- [Background] Andrews B, Wilding JM. The relation of depression and anxiety to life-stress and achievement in students. Br J Psychol. 2004 Nov;95(Pt 4):509-21. doi: 10.1348/0007126042369802. PMID 15527535
- [Background] Kajitani K, Higashijima I, Kaneko K, Matsushita T, Fukumori H, Kim D. Short-term effect of a smartphone application on the mental health of university students: A pilot study using a user-centered design self-monitoring application for mental health. PLoS One. 2020 Sep 25;15(9):e0239592. doi: 10.1371/journal.pone.0239592. eCollection 2020. PMID 32976515
- [Background] Musiat P, Conrod P, Treasure J, Tylee A, Williams C, Schmidt U. Targeted prevention of common mental health disorders in university students: randomised controlled trial of a transdiagnostic trait-focused web-based intervention. PLoS One. 2014 Apr 15;9(4):e93621. doi: 10.1371/journal.pone.0093621. eCollection 2014. PMID 24736388
- [Background] Huberty J, Green J, Glissmann C, Larkey L, Puzia M, Lee C. Efficacy of the Mindfulness Meditation Mobile App "Calm" to Reduce Stress Among College Students: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Jun 25;7(6):e14273. doi: 10.2196/14273. PMID 31237569
- [Background] Aboalshamat K, Hou XY, Strodl E. The impact of a self-development coaching programme on medical and dental students' psychological health and academic performance: a randomised controlled trial. BMC Med Educ. 2015 Aug 19;15:134. doi: 10.1186/s12909-015-0412-4. PMID 26286331
- [Background] Gopalakrishnan V, Umabalan T, Affan M, Zamri AA, Kamal A, Sandheep S. Stress perceived by houseman in a hospital in northern Malaysia. Med J Malaysia. 2016 Feb;71(1):8-11. PMID 27130736
- [Background] Yeoh CM, Thong KS, Seed HF, Nur Iwana AT, Maruzairi H. Psychological morbidities amongst house officers in Sarawak General Hospital Kuching. Med J Malaysia. 2019 Aug;74(4):307-311. PMID 31424038
- [Background] Rashid AA, Ghazali SS, Mohamad I, Mawardi M, Musa H, Roslan D. The effectiveness of a Malaysian House Officer (HO) preparatory course for medical graduates on self-perceived confidence and readiness: A quasi-experimental study. PLoS One. 2020 Jul 17;15(7):e0235685. doi: 10.1371/journal.pone.0235685. eCollection 2020. PMID 32678838
- [Derived] Lim YS, Quek JH, Ching XW, Lim DTR, Lim KG, Thuraisingham C, George PP. Efficacy of a Text-Based Mental Health Coaching App in Improving the Symptoms of Stress, Anxiety, and Depression: Randomized Controlled Trial. JMIR Form Res. 2023 Sep 22;7:e46458. doi: 10.2196/46458. PMID 37738081
- See also: The Burden of Mental Illness: An Emerging Global Disaster. Sungai Buloh — https://jchs-medicine.uitm.edu.my/images/manuscript/vol3issue1/review/p5-12/The-Burden-of-Mental-Illness-An-Emerging-Global-Disaster.pdf
- See also: Malaysian Healthcare Performance Unit, Malaysian Healthcare Performance: Technical Report 2016, Ministry of Health Malaysia, Putrajaya — https://www.moh.gov.my/moh/resources/Penerbitan/Laporan/Umum/Mental%20Healthcare%20Performance%20Report%202016.pdf
- See also: Information about Mental Illness and the Brain. — https://www.ncbi.nlm.nih.gov/books/NBK20369/
- See also: Common Mental Health Disorders: Identification and Pathways to Care. — https://www.ncbi.nlm.nih.gov/books/NBK92254/
- See also: A qualitative exploration of the perspectives of mental health professionals on stigma and discrimination of mental illness in Malaysia. Int J Ment Health Syst 9, 10 (2015). — https://doi.org/10.1186/s13033-015-0002-1
- See also: Mental Health of the world — http://OurWorldInData.org.
- See also: Mental Health and Coping Response among Malaysian Adults during COVID-19 Pandemic Movement Control Order — http://www.jcreview.com/?mno=45437
- See also: The APEC Digital Hub-WONCA Collaborative Framework on Integration of Mental Health into Primary Care in the Asia Pacific — https://doi.org/10.2147/JMDH.S271070
- See also: Resilience: A definition in context. Australian Community Psychologist — https://www.psychology.org.au/APS/media/ACP/ACP-1-2010.pdf
- See also: Building your resilience — https://www.apa.org/topics/resilience
- See also: The Prevalence and Associated Factors of Depression, Anxiety and Stress of First Year Undergraduate Students in a Public Higher Learning Institution in Malaysia. — https://link.springer.com/article/10.1007/s10826-019-01537-y
- See also: Stress among Medical Students and Its Association with Substance Use and Academic Performance — https://www.researchgate.net/publication/285657055_Stress_among_Medical_Students_and_Its_Association_with_Substance_Use_and_Academic_Performance
- See also: The challenges and mental health issues of academic trainees. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7199285/
- See also: The Global Prevalence of Anxiety Among Medical Students: A Meta-Analysis — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6696211/
- See also: National Centre for Education Statistics. Nontraditional Undergraduates / Definitions and Data — https://nces.ed.gov/pubs/web/97578e.asp
- See also: Life satisfaction among university students in a Canadian Prairie City: a multivariate analysis — https://link.springer.com/article/10.1007/s11205-004-7526-0
- See also: Doctors still see own mental health problems as sign of weakness, research finds — https://www.bmj.com/content/365/bmj.l1861.full
- See also: Road to resilience: a systematic review and meta-analysis of resilience training programmes and interventions — https://bmjopen.bmj.com/content/8/6/e017858
- See also: Coping Skills and Burnout among Medical Officers in a Malaysian Tertiary Hospital — http://ir.uitm.edu.my/id/eprint/29899/1/AJ_NUR%20FAIZAH%20ALI%20AJE-BS%20B%2020.pdf
- See also: A Study of BetterHelp Text-Based Counseling — https://assets.betterhelp.com/research/Study_of_BetterHelp_Text-Based_Counseling.pdf
- See also: Application of Synchronous Text-Based Dialogue Systems in Mental Health Interventions: Systematic Review — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5595406/
- See also: Two-way messaging therapy for depression and anxiety: longitudinal response trajectories — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7291694/
- See also: Impact of a mobile phone and web program on symptom and functional outcomes for people with mild-to-moderate depression, anxiety and stress: a randomised controlled trial — https://link.springer.com/article/10.1186/1471-244X-13-312#citeas
- See also: An Empathy-Driven, Conversational Artificial Intelligence Agent (Wysa) for Digital Mental Well-Being: Real-World Data Evaluation Mixed-Methods Study — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6286427/
- See also: Long-Term Outcomes of a Therapist-Supported, Smartphone-Based Intervention for Elevated Symptoms of Depression and Anxiety: Quasiexperimental, Pre-Postintervention Study — https://mhealth.jmir.org/2019/8/e14284/